CLINICAL TRIAL: NCT00001402
Title: Assessment of Metabolic Function and Perfusion Using Positron Emission Tomography: An Analysis of Patients With Congestive Cardiomyopathy Before and After Beta-Blockers
Brief Title: PET Scan to Determine Areas of Blood Flow and Activity in the Hearts of Patients With Heart Disease Taking Beta-Blockers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 940054; 94-H-0054
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-12

CONDITIONS: Heart Failure, Congestive
Keywords: Dilated Cardiomyopathy; Hibernating Myocardium; Ischemic Cardiomyopathy; Metoprolol; Stress Thallium Scintigraphy; Congestive Cardiomyopathy; Congestive Heart Failure; Heart Failure
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated | interventions — Positron-Emission Tomography

INTERVENTIONS:
Device: PET scan

SUMMARY:
The human heart is divided into four chambers. One of the four chambers, the left ventricle, is the chamber mainly responsible for pumping blood out of the heart into the circulation. Diseases of the heart like congestive heart failure (CHF), can cause the left ventricle to function improperly.

Medications called beta-blockers appear to reverse the abnormalities in the left ventricle and frequently improve the function of the left ventricle in patients with different kinds of heart disease. How beta-blockers improve left ventricle function is unknown.

One possible reason for improved function of the left ventricle with beta-blockers is improved blood flow to the heart muscle. When a region of the heart is active, it uses more fuel in the form of oxygen and sugar (glucose). As heart activity increases, blood flow to and from the area of activity increases also. Knowing these facts, researchers can use radioactive sugar (glucose) and positron emission tomography (PET) scans to observe what areas of the heart are receiving more blood flow.

In this study researchers plan to measure glucose use in heart muscle and blood flow to the heart muscle in patients with CHF taking beta-blockers.

DETAILED DESCRIPTION:
Deterioration in left ventricular function, which is characteristic in patients with congestive heart failure, appears to be a multifactorial process. Beta-blockers appear to reverse the deterioration and frequently improve left ventricular function in patients with both ischemic and non-ischemic cardiomyopathies. The mechanism by which beta-blockers improve ejection fraction is not known. Although it is well established that regional flow, function and metabolism may improve after coronary revascularization whether beta-blocker therapy will have similar salutary results in patients with congestive heart failure is unknown. The aim of this study is to: 1) quantitate regional glucose uptake and regional blood flow before and after chronic beta-blocker administration to patients with congestive heart failure using positron emission tomography, 2) determine if alteration in either regional glucose or lipid uptake or regional blood flow correlate with improvement in wall motion and global left ventricular function, and 3) determine if ischemic and nonischemic myocardium differ in blood flow or metabolism.

ELIGIBILITY:
Left ventricular ejection fraction by radionuclide angiography of less than or equal to 40%.

New York Heart Association class II, III or IV symptoms on standard heart failure medications which my include digoxin, diuretics and angiotensin converting enzyme inhibitors for at least one month prior to enrollment.

Ischemic cardiomyopathy if enzymes document an MI or 70% or greater stenosis in one major vessel.

Dilated cardiomyopathy-if no coronary disease.

No pregnant or lactating women.

No women of child-bearing age not on proven birth control.

No severe hepatic or renal disease.

No diabetes mellitus or fasting glucose greater than or equal to 120 mg/dl.

No primary valvular heart disease.

No PTCA or CABG within 3 months of enrollment.

No history of myocardial infarction or unstable angina within past 2 months.

No resting heart rate less than 60 bpm.

No A-V block greater than 1 degree block without pacemaker.

No severe ETOH abuse within 6 months of enrollment.

No severe bronchospasm.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130
Dates: Start 1994-01; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Eichhorn EJ, Heesch CM, Barnett JH, Alvarez LG, Fass SM, Grayburn PA, Hatfield BA, Marcoux LG, Malloy CR. Effect of metoprolol on myocardial function and energetics in patients with nonischemic dilated cardiomyopathy: a randomized, double-blind, placebo-controlled study. J Am Coll Cardiol. 1994 Nov 1;24(5):1310-20. doi: 10.1016/0735-1097(94)90114-7. PMID 7930255
- [Background] Kjekshus JK, Mjos OD. Effect of free fatty acids on myocardial function and metabolism in the ischemic dog heart. J Clin Invest. 1972 Jul;51(7):1767-76. doi: 10.1172/JCI106978. PMID 5032525